CLINICAL TRIAL: NCT02428712
Title: A Phase 1/2a Study to Assess the Safety, Pharmacokinetics, and Pharmacodynamics of FORE8394 in Patients With Advanced Unresectable Solid Tumors
Brief Title: A Study of FORE8394 as a Single Agent in Patients With Advanced Unresectable Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fore Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLX120-03
Record Dates: First submitted 2015-04-20; First posted 2015-04-29 (Estimated); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Advanced Unresectable Solid Tumors; BRAF-mutated Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FORE8394 (Experimental): Group A: Phase 1-Dose Escalation: Adult patients.
  Group B: Phase 1-Dose Escalation: Pediatric patients.
  Phase 2a-Dose Extension: Adult patients with advanced unresectable solid tumors will be enrolled among two cohorts.
  * Cohort 1: Activating BRAF V600 mutations (glioma patients only)
  * Cohort 2: Activating BRAF non-V600 mutations
  Phase 2a-RP2D Confirmation: Adult patients.
  Phase 2a-RP2D Redefinition and Extension:
  * Cohort 3: Activating BRAF V600 or activating non-V600 mutation
  * Cohort 4: Activating BRAF non-V600 mutations
  Phase 2a-RP2D Redefinition:
  * Cohort 6A: Advanced activating BRAF-mutated solid tumors
  * Cohort 7A: Advanced activating BRAF-mutated solid tumors
  * Cohort 8A: Advanced activating BRAF-mutated solid tumors
  Interventions: Drug: FORE8394

INTERVENTIONS:
Drug: FORE8394

SUMMARY:
The objective of this study is to determine the safety, pharmacokinetics, maximum tolerated dose/recommended Phase 2 dose, and efficacy of FORE8394.

DETAILED DESCRIPTION:
Dose Escalation (Part 1): To evaluate safety, pharmacokinetics, pharmacodynamics of FORE8394 in adult and pediatric patients with advanced BRAF- mutated tumors, and to identify the recommended Phase 2 Dose.

Dose Extension (Part 2): To access objective tumor response to FORE8394 treatment in adult and in adolescent patients with advanced BRAF- mutated tumors, to access RECIST, and to access pharmacokinetics, pharmacodynamics, and safety.

ELIGIBILITY:
Inclusion Criteria- Group A:

* Age ≥ 10 years and at least 30 kg.
* Phase 1-Dose Escalation (no longer enrolling as of Protocol Amendment 10): Patients with histologically confirmed advanced solid tumors who are refractory to, relapsed after, or intolerant to standard therapy or for whom no standard therapy exists.
* Phase 2a-Dose Extension: Criteria for Dose Extension [HME] Cohort 1 or Cohort 2, are specified below:

  * Phase 2a-Dose Extension-Cohort 1

    1. Patients with solid tumors (as of Amendment 10, only subjects with glioma tumors) driven by an activating BRAF-V600 mutation
    2. Patients with no prior exposure to BRAF-directed therapy and for whom no standard therapy exists.
  * Phase 2a-Dose Extension-Cohort 2

    1. Patients with solid tumors driven by an activating BRAF non-V600 mutation, which can include a point mutation, gene amplification, fusion, insertion, or deletion
    2. Participants with no prior exposure to BRAF-directed therapy and for whom no standard therapy exists.
* Phase 2a - RP2D Redefinition Extension: Following RP2D redefinition, extension participants must meet criteria for Cohort 3 or Cohort 4 as specified below:

  1. Cohort 3: Participants with advanced unresectable gliomas driven by an activating BRAF V600 or activating non-V600 mutation who have no prior exposure to a BRAF, MEK, or ERK inhibitor and for whom no standard therapy exists.
  2. Cohorts 4-8: Participants with advanced solid tumors driven by activating BRAF non V600 mutations, which can include a point mutation, gene amplification, fusion, insertion, deletion, or alternative splicing, who have no prior exposure to a BRAF, MEK, or ERK inhibitor.
* Measurable disease by RECIST 1.1.
* RANOS (CNS tumors) - High Grade Glioma for high grade glioma (Grades 3 and 4) and RANO-Low Grade Glioma for low grade glioma.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Adequate hematologic, hepatic, and renal function.
* Women of child-bearing potential must have a negative pregnancy test and must agree to use an effective form of contraception from the time of the negative pregnancy test up to 3 months after the last dose of study drug. Women of non-child-bearing potential may be included if they are either surgically sterile or have been postmenopausal for ≥ 1 year.
* Fertile men must agree to use an effective method of birth control during the study and for up to 3 months after the last dose of study drug.
* Completion of previous anti-cancer therapy at least 2 weeks before study drug initiation.

Exclusion Criteria- Group A:

* Participants with known co-occurring RAS-related mutations or RTK activation are not allowed.
* Major surgical procedure, open biopsy (excluding skin cancer resection), or significant traumatic injury within 14 days of initiating study drug or anticipation of the need for major surgery during the study.
* Uncontrolled intercurrent illness.
* Patients with colorectal cancer or pancreatic cancer
* Active secondary malignancy unless the malignancy is not expected to interfere with the evaluation of safety and is approved by the Medical Monitor. Patients with a completely treated prior malignancy and no evidence of disease for ≥ 2 years are eligible.
* Refractory nausea and vomiting, malabsorption, external biliary shunt, or significant bowel resection that would preclude adequate absorption.
* Clinically significant cardiac disease.
* Known infection with HIV, HBV, or HCV or a known carrier of HBV or HCV.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2024-07-12 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) of FORE8394 | First dose of FORE8394 up to 30 days after end of treatment
Maximum concentration (Cmax) of FORE8394 | First dose of FORE8394 up to 30 days after end of treatment
Time to peak concentration (Tmax) of FORE8394 | First dose of FORE8394 up to 30 days after end of treatment
Half life (T1/2) of FORE8394 | First dose of FORE8394 up to 30 days after end of treatment
Number of participants with Treatment Emergent Adverse Events (TEAEs) as assessed by CTCAE v4.0. | First dose of FORE8394 up to 30 days after end of treatment
To identify the recommended Phase 2 dose (RP2D) of FORE8394 in Group A (adult patients) for further evaluation in Dose Extension. | 2 years
Compare AUC of FORE8394 with FORE8394 | First dose of FORE8394 up to 30 days after end of treatment
Compare Cmax of FORE8394 with FORE8394 | First dose of FORE8394 up to 30 days after end of treatment
Compare Tmax of FORE8394 with FORE8394 | First dose of FORE8394 up to 30 days after end of treatment
Compare T1/2 of FORE8394 with FORE8394 | First dose of FORE8394 up to 30 days after end of treatment
To determine the overall response rate of FORE8394 treatment at the applicable RP2D in a) Group A, Cohort 1, and b) Group A, Cohort 2. | 5 years

SECONDARY OUTCOMES:
To evaluate the duration of response (defined as time of initial response to progressive disease or death) at the applicable RP2D in Dose Extension. | 5 years
To evaluate the progression free survival (defined as time of first dose to progressive disease or death) at the applicable RP2D in Dose Extension. | 5 years
Clinical benefit rate (defined as stable disease, partial response and complete response) after 24 weeks on study | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Stacie Peacock Shepherd, MD, PhD, Study Chair — Fore Biotherapeutics U.S. Inc.
Locations (13):
- United States (13):
  - HonorHealth, Scottsdale, Arizona
  - St. Joseph's Hospital at Orange, Orange, California
  - Stanford Hospitals and Clinics, Stanford, California
  - University of Miami, Miami, Florida
  - Community Health Network, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Capital Regional Medical Center, Jefferson City, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Baptist Cancer Center, Memphis, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Children's Hospital (Baylor College of Medicine), Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah